CLINICAL TRIAL: NCT01546922
Title: A Randomized Double Blind Cross-over Study of the Effects of Low Dose and High Dose Hydrocortisone Replacement Therapy on Cognition, Quality of Life, Metabolic Profile and Somatosensation in Patients With Secondary Adrenal Insufficiency
Brief Title: Hydrocortisone Replacement in Patients With Secondary Adrenal Insufficiency (SUPREME CORT)
Acronym: SUPREME CORT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, A.P. van Beek, MD PhD, Principal Investigator, University Medical Center Groningen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NL 35668.042.11; 2011-000864-82 (EudraCT Number)
Record Dates: First submitted 2012-02-07; First posted 2012-03-07 (Estimated); Results first posted 2014-07-14 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-06

CONDITIONS: Adrenal Insufficiency
Keywords: Hydrocortisone; Cognition; Adrenal insufficiency; Quality of Life; Common Somatic Complaints; Cardiovascular/Metabolic Profile; Somatosensation
MeSH Terms: conditions — Adrenal Insufficiency | interventions — Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- First low dose HC followed by high dose HC (Active Comparator): First low dose of hydrocortisone = 0.2-0.3 mg/kg body weight for 10 weeks followed by a high dose of hydrocortisone = 0.4-0.6 mg/kg body weight
  Interventions: Drug: Hydrocortisone
- First high dose HC followed by low dose HC (Active Comparator): First a high dose of hydrocortisone = 0.4-0.6 mg/kg body weight for 10 weeks followed by a low dose of hydrocortisone = 0.2-0.3 mg/kg body weight
  Interventions: Drug: Hydrocortisone

INTERVENTIONS:
Drug: Hydrocortisone — Patients receive either a low dose HC (0.2-0.3 mg/kg body weight) for 10 weeks followed by 10 weeks of high dose HC (0.4-0.6 mg/kg body weight) or vice versa.

SUMMARY:
The aim of this study is to investigate whether a physiologically low hydrocortisone (HC) dose is better for cognition as compared to a physiologically high HC dose. In addition, quality of life, metabolic profile and somatosensation will be described in relation to HC dose.

DETAILED DESCRIPTION:
* Rationale: A wide variety in hydrocortisone (HC) substitution dose-regimens are considered physiological for patients with adrenal insufficiency. However, it is likely that cognition is negatively influenced by higher cortisol exposure to the brain. No studies have been performed to assess the effects of treatment regimens with a low physiological HC substitution dose on cognition in comparison to a high physiological HC substitution dose. These treatment regimens should take body weight and multiple dosing into account. In addition, substitution doses should be monitored by clinical evaluation and biochemical analysis for adverse effects associated with over- or under-replacement.
* Intervention: Patients with secondary adrenal insufficiency will be randomized in two groups to receive either a low dose HC (0.2-0.3 mg/kg body weight) for 10 weeks followed by 10 weeks of high dose HC (0.4-0.6 mg/kg body weight) or vice versa. At baseline and after both treatment periods, patients will be tested.

ELIGIBILITY:
Inclusion Criteria:

* Patients with secondary adrenal insufficiency.
* Age ≥ 18 - 75 years
* ≥ One year after tumor treatment with surgery and/or radiotherapy
* On stable concomitant medications for at least six months prior to entry of study
* Body weight 50-100 kg

Exclusion Criteria:

* Inability of legal consent
* Documented cognitive impairment
* Drug abuse/dependence
* History of / current psychiatric disorders
* Use of anti-epileptics (e.g. carbamezapine)
* Cushing Disease
* Type 1 diabetes or Type 2 diabetes with medication known to induce hypoglycemia (f.e. Sulfonylurea derivatives
* Current treatment for second malignancy
* Have a significant medical condition (e.g. hepatic, respiratory, or cardiovascular) which, in the opinion of the investigator, may interfere with the interpretation of results and safety or efficacy evaluations.
* A history of frequent hypocortisolism
* Hospitalization during study
* Work in shifts

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2012-02; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: André P van Beek, Dr., Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Centre Groningen, Groningen, Provincie Groningen, Netherlands

REFERENCES:
- [Derived] Sorgdrager FJH, Werumeus Buning J, Bos EH, Van Beek AP, Kema IP. Hydrocortisone Affects Fatigue and Physical Functioning Through Metabolism of Tryptophan: A Randomized Controlled Trial. J Clin Endocrinol Metab. 2018 Sep 1;103(9):3411-3419. doi: 10.1210/jc.2018-00582. PMID 29982583
- [Derived] Werumeus Buning J, Touw DJ, Brummelman P, Dullaart RPF, van den Berg G, van der Klauw MM, Kamp J, Wolffenbuttel BHR, van Beek AP. Pharmacokinetics of oral hydrocortisone - Results and implications from a randomized controlled trial. Metabolism. 2017 Jun;71:7-16. doi: 10.1016/j.metabol.2017.02.005. Epub 2017 Feb 13. PMID 28521880
- [Derived] Werumeus Buning J, van Faassen M, Brummelman P, Dullaart RP, van den Berg G, van der Klauw MM, Kerstens MN, Stegeman CA, Muller Kobold AC, Kema IP, Wolffenbuttel BH, van Beek AP. Effects of Hydrocortisone on the Regulation of Blood Pressure: Results From a Randomized Controlled Trial. J Clin Endocrinol Metab. 2016 Oct;101(10):3691-3699. doi: 10.1210/jc.2016-2216. Epub 2016 Aug 4. PMID 27490921
- [Derived] Werumeus Buning J, Brummelman P, Koerts J, Dullaart RP, van den Berg G, van der Klauw MM, Sluiter WJ, Tucha O, Wolffenbuttel BH, van Beek AP. Hydrocortisone Dose Influences Pain, Depressive Symptoms and Perceived Health in Adrenal Insufficiency: A Randomized Controlled Trial. Neuroendocrinology. 2016;103(6):771-8. doi: 10.1159/000442985. Epub 2015 Dec 9. PMID 26646751
- [Derived] Werumeus Buning J, Brummelman P, Koerts J, Dullaart RP, van den Berg G, van der Klauw MM, Tucha O, Wolffenbuttel BH, van Beek AP. The effects of two different doses of hydrocortisone on cognition in patients with secondary adrenal insufficiency--results from a randomized controlled trial. Psychoneuroendocrinology. 2015 May;55:36-47. doi: 10.1016/j.psyneuen.2015.02.001. Epub 2015 Feb 10. PMID 25705800

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Sixty-three patients were included in the study. Three patients withdrew from the study during the run-in phase, therefore a total of 60 patients started the first treatment period.
Groups:
- First a Low Dose of HC Followed by a High Dose of HC: First low dose of hydrocortisone = 0.2-0.3 mg/kg body weight for 10 weeks followed by a high dose of hydrocortisone = 0.4-0.6 mg/kg body weight
- First a High Dose of HC Followed by a Low Dose of HC: First high dose of hydrocortisone = 0.4-0.6 mg/kg body weight for 10 weeks followed by a low dose of hydrocortisone = 0.2-0.3 mg/kg body weight
Period: First Period of 10 Weeks
Arm/Group | First a Low Dose of HC Followed by a High Dose of HC | First a High Dose of HC Followed by a Low Dose of HC
Started | 30 | 30
Completed | 25 | 28
Not Completed | 5 | 2
Not completed — Protocol Violation | 3 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Investigator's judgment | 1 | 0
Period: Second Period of 10 Weeks
Arm/Group | First a Low Dose of HC Followed by a High Dose of HC | First a High Dose of HC Followed by a Low Dose of HC
Started | 25 | 28
Completed | 22 | 25
Not Completed | 3 | 3
Not completed — Protocol Violation | 3 | 1
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Population: The 47 participants completing both study periods were used for further analysis.
Groups:
- All Participants: All participants completing both study periods
Arm/Group | All Participants
Number analyzed (Participants) | 47
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 55 (14) [43 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 29
Region of Enrollment [Number; unit: participants]
  Netherlands | 47
Age at diagnosis [Median (Inter-Quartile Range); unit: years] | 31 (16) [20 to 46]
Childhood onset/Adult onset [Number; unit: participants]
  Childhood onset | 6
  Adult onset | 41
Body weight [Median (Inter-Quartile Range); unit: kilogram] | 82.5 (13.9) [72.2 to 93.0]
Type of surgery [Number; unit: participants] — A total of 32 participants underwent surgery
  participants
    Transsphenoïdal surgery | 23
    Craniotomy | 9
Age at surgery [Median (Inter-Quartile Range); unit: years] | 39 [28 to 50]
Median time since surgery [Median (Inter-Quartile Range); unit: years] | 11 [6 to 20]
Patients with a second surgery [Number; unit: participants] | 5
Type of radiotherapy [Number; unit: participants] — A total of 19 participants received radiotherapy
  participants
    Pituitary radiotherapy | 16
    Cranial irradiation | 2
    Radiotherapy for extracranial tumors | 1
Age at radiotherapy [Median (Inter-Quartile Range); unit: years] | 43 [25 to 52]
Median time since radiotherapy [Median (Inter-Quartile Range); unit: years] | 12 [9 to 22]
Total daily dose hydrocortisone treatment prior to randomization [Median (Inter-Quartile Range); unit: mg/day] | 25 [20 to 30]
Dose per kg body weight prior to randomization [Median (Inter-Quartile Range); unit: mg/kg body weight] | 0.32 [0.25 to 0.35]
Number of daily dosings prior to randomization [Number; unit: participants]
  1 dose per day | 3
  2 doses per day | 33
  3 doses per day | 11
Duration of hydrocortisone treatment prior to randomization [Median (Inter-Quartile Range); unit: years] | 12 [5 to 22]
Number of hormonal replacements [Number; unit: participants]
  1 hormonal replacement | 3
  2 hormonal replacements | 9
  3 hormonal replacements | 21
  4 hormonal replacements | 11
  5 hormonal replacements | 3
Thyroid hormone substitution [Number; unit: participants] | 43
Growth hormone (GH) [Number; unit: participants]
  Participants substituted | 21
  Participants unsubstituted | 10
Sex hormone [Number; unit: participants]
  Participants substituted | 27
  Men: testosterone substitution | 23
  Premenopausal women: estrogen substitution | 4
Desmopressin substitution [Number; unit: participants] | 9

OUTCOME MEASURES:

1. Primary Outcome: Change in Cognition After 10 Weeks of Treatment With a Low Dose of Hydrocortisone Compared to 10 Weeks of Treatment With a High Dose of Hydrocortisone.
Description: Cognitive domains to be tested: memory, executive functioning, attention and social cognition.
  The psychological tests consist of oral and written questions or computer tasks.
  Data is given as Z-scores based on normative data. Higher Z-scores represent a better performance.
Time Frame: After completion of treatment period 1 (that is after 10 weeks from baseline) and after treatment period 2 (that is after 20 weeks from baseline).
Population: The participants completing both study periods were analyzed
Measure: Mean (Standard Deviation); unit: Z-scores based on normative data.
Groups:
- Low Dose of Hydrocortisone: Results from the participants while receiving the low dose of hydrocortisone
- High Dose of Hydrocortisone: Results from the participants while receiving the high dose of hydrocortisone
Arm/Group | Low Dose of Hydrocortisone | High Dose of Hydrocortisone
Number analyzed (Participants) | 47 | 47
Z-scores based on normative data.
  RBMT-Immediate Memory | -0.41 (0.95) | -0.42 (1.33)
  RBMT-Delayed Memory | 0.07 (0.98) | 0.10 (1.33)
  RBMT-Delayed corrected for immediate memory | 0.85 (1.09) | 0.89 (1.34)
  15 Words Test-Short-term memory | 0.36 (1.01) | -0.03 (1.03)
  15 Words Test-Total immediate memory | 0.43 (1.02) | 0.25 (0.92)
  15 Words Test - Learning Score | 0.08 (1.05) | 0.38 (1.19)
  15 Words Test - Delayed Memory | 0.02 (1.04) | 0.23 (0.97)
  15 Words Test - Delayed corrected for total memory | -0.30 (0.99) | -0.16 (0.99)
  15 Words Test-Recognition | -0.11 (0.88) | 0.08 (0.71)
  Digit Span forward - Short term memory | 0.49 (0.97) | 0.56 (0.97)
  Rey Complex Figure - Immediate memory | 1.14 (1.26) | 1.40 (1.29)
  Rey Complex Figure - Delayed memory | 1.11 (1.22) | 1.28 (1.29)
  Divided attention-reaction time auditory response | -0.87 (0.81) | -0.89 (0.82)
  Divided attention-reaction time visual response | -0.06 (1.00) | 0.03 (0.94)
  Divided attention - Number of omission errors | -0.02 (0.86) | -0.14 (0.93)
  Divided attention - Number of commission errors | 0.30 (1.01) | 0.34 (0.76)
  Visual scanning - Reaction time for target stimuli | -0.38 (1.04) | -0.36 (1.03)
  Visual scanning - Number of omission errors | -0.03 (1.06) | 0.08 (1.08)
  Visual scanning - Number of commission errors | -0.72 (0.26) | -0.70 (0.28)
  Alertness - Reaction time tonic alertness | -0.90 (0.73) | -0.99 (0.73)
  Alertness - Reaction time phasic alertness | -1.03 (0.67) | -1.10 (0.66)
  Semantic fluency | 0.02 (1.24) | 0.09 (1.18)
  Phonemic fluency | 0.32 (1.48) | 0.21 (1.31)
  Digit Span backwards-Working memory | 0.05 (0.86) | -0.01 (1.02)
  Trail Making Test - Time condition A | -0.32 (1.14) | -0.26 (1.06)
  Trail Making Test - Time condition B | 0.16 (1.46) | 0.18 (1.31)
  Trail Making Test - Condition B/A | 0.37 (1.42) | 0.36 (1.48)
  Social Cognition | -0.67 (1.20) | -0.71 (1.15)
Statistical Analysis 1: Comparison: Low Dose of Hydrocortisone vs High Dose of Hydrocortisone; Rivermead Behavioural Memory Test (RBMT) - Immediate memory; Test type: Superiority or Other; p = 0.861, Wilcoxon (Mann-Whitney) — A Bonferroni correction for multiple comparisons was applied, resulting in a significance level of 0.001
Statistical Analysis 2: Comparison: Low Dose of Hydrocortisone vs High Dose of Hydrocortisone; RBMT - Delayed memory; Test type: Superiority or Other; p = 0.668, Wilcoxon (Mann-Whitney) — A Bonferroni correction for multiple comparisons was applied, resulting in a significance level of 0.001
Statistical Analysis 3: Comparison: Low Dose of Hydrocortisone vs High Dose of Hydrocortisone; RBMT-Delayed corrected for immediate memory; Test type: Superiority or Other; p = 0.713, Wilcoxon (Mann-Whitney) — A Bonferroni correction for multiple comparisons was applied, resulting in a significance level of 0.001
Statistical Analysis 4: Comparison: Low Dose of Hydrocortisone vs High Dose of Hydrocortisone; 15 Words Test - Short-term memory; Test type: Superiority or Other; p = 0.028, Wilcoxon (Mann-Whitney) — A Bonferroni correction for multiple comparisons was applied, resulting in a significance level of 0.001
Statistical Analysis 5: Comparison: Low Dose of Hydrocortisone vs High Dose of Hydrocortisone; 15 Words Test - Total immediate memory; Test type: Superiority or Other; p = 0.227, Wilcoxon (Mann-Whitney) — A Bonferroni correction for multiple comparisons was applied, resulting in a significance level of 0.001
Statistical Analysis 6: Comparison: Low Dose of Hydrocortisone vs High Dose of Hydrocortisone; 15 Words Test - Learning Score; Test type: Superiority or Other; p = 0.130, Wilcoxon (Mann-Whitney) — A Bonferroni correction for multiple comparisons was applied, resulting in a significance level of 0.001
Statistical Analysis 7: Comparison: Low Dose of Hydrocortisone vs High Dose of Hydrocortisone; 15 Words Test- Delayed memory; Test type: Superiority or Other; p = 0.106, Wilcoxon (Mann-Whitney) — A Bonferroni correction for multiple comparisons was applied, resulting in a significance level of 0.001
Statistical Analysis 8: Comparison: Low Dose of Hydrocortisone vs High Dose of Hydrocortisone; 15 Words Test - Delayed corrected for total memory; Test type: Superiority or Other; p = 0.350, Wilcoxon (Mann-Whitney) — A Bonferroni correction for multiple comparisons was applied, resulting in a significance level of 0.001
Statistical Analysis 9: Comparison: Low Dose of Hydrocortisone vs High Dose of Hydrocortisone; 15 Words Test - Recognition; Test type: Superiority or Other; p = 0.093, Wilcoxon (Mann-Whitney) — A Bonferroni correction for multiple comparisons was applied, resulting in a significance level of 0.001
Statistical Analysis 10: Comparison: Low Dose of Hydrocortisone vs High Dose of Hydrocortisone; Digit Span forward - Short-term memory; Test type: Superiority or Other; p = 0.614, Wilcoxon (Mann-Whitney) — A Bonferroni correction for multiple comparisons was applied, resulting in a significance level of 0.001
Statistical Analysis 11: Comparison: Low Dose of Hydrocortisone vs High Dose of Hydrocortisone; Rey Complex Figure - Immediate memory; Test type: Superiority or Other; p = 0.111, Wilcoxon (Mann-Whitney) — A Bonferroni correction for multiple comparisons was applied, resulting in a significance level of 0.001
Statistical Analysis 12: Comparison: Low Dose of Hydrocortisone vs High Dose of Hydrocortisone; Rey Complex Figure - Delayed memory; Test type: Superiority or Other; p = 0.451, Wilcoxon (Mann-Whitney) — A Bonferroni correction for multiple comparisons was applied, resulting in a significance level of 0.001
Statistical Analysis 13: Comparison: Low Dose of Hydrocortisone vs High Dose of Hydrocortisone; Divided attention-Reaction time auditory response; Test type: Superiority or Other; p = 0.905, Wilcoxon (Mann-Whitney) — A Bonferroni correction for multiple comparisons was applied, resulting in a significance level of 0.001
Statistical Analysis 14: Comparison: Low Dose of Hydrocortisone vs High Dose of Hydrocortisone; Divided attention-Reaction time visual response; Test type: Superiority or Other; p = 0.502, Wilcoxon (Mann-Whitney) — A Bonferroni correction for multiple comparisons was applied, resulting in a significance level of 0.001
Statistical Analysis 15: Comparison: Low Dose of Hydrocortisone vs High Dose of Hydrocortisone; Divided attention-Number of omission errors; Test type: Superiority or Other; p = 0.531, Wilcoxon (Mann-Whitney) — A Bonferroni correction for multiple comparisons was applied, resulting in a significance level of 0.001
Statistical Analysis 16: Comparison: Low Dose of Hydrocortisone vs High Dose of Hydrocortisone; Divided attention-Number of commission errors; Test type: Superiority or Other; p = 0.681, Wilcoxon (Mann-Whitney) — A Bonferroni correction for multiple comparisons was applied, resulting in a significance level of 0.001
Statistical Analysis 17: Comparison: Low Dose of Hydrocortisone vs High Dose of Hydrocortisone; Visual scanning - Reaction time for target stimuli; Test type: Superiority or Other; p = 0.713, Wilcoxon (Mann-Whitney) — A Bonferroni correction for multiple comparisons was applied, resulting in a significance level of 0.001
Statistical Analysis 18: Comparison: Low Dose of Hydrocortisone vs High Dose of Hydrocortisone; Visual scanning - Number of omission errors; Test type: Superiority or Other; p = 0.229, Wilcoxon (Mann-Whitney) — A Bonferroni correction for multiple comparisons was applied, resulting in a significance level of 0.001
Statistical Analysis 19: Comparison: Low Dose of Hydrocortisone vs High Dose of Hydrocortisone; Visual scanning - Number of commission errors; Test type: Superiority or Other; p = 0.329, Wilcoxon (Mann-Whitney) — A Bonferroni correction for multiple comparisons was applied, resulting in a significance level of 0.001
Statistical Analysis 20: Comparison: Low Dose of Hydrocortisone vs High Dose of Hydrocortisone; Alertness - Reaction time tonic alertness; Test type: Superiority or Other; p = 0.192, Wilcoxon (Mann-Whitney) — A Bonferroni correction for multiple comparisons was applied, resulting in a significance level of 0.001
Statistical Analysis 21: Comparison: Low Dose of Hydrocortisone vs High Dose of Hydrocortisone; Alertness - Reaction time phasic alertness; Test type: Superiority or Other; p = 0.164, Wilcoxon (Mann-Whitney) — A Bonferroni correction for multiple comparisons was applied, resulting in a significance level of 0.001
Statistical Analysis 22: Comparison: Low Dose of Hydrocortisone vs High Dose of Hydrocortisone; Semantic fluency; Test type: Superiority or Other; p = 0.536, Wilcoxon (Mann-Whitney) — A Bonferroni correction for multiple comparisons was applied, resulting in a significance level of 0.001
Statistical Analysis 23: Comparison: Low Dose of Hydrocortisone vs High Dose of Hydrocortisone; Phonemic fluency; Test type: Superiority or Other; p = 0.572, Wilcoxon (Mann-Whitney) — A Bonferroni correction for multiple comparisons was applied, resulting in a significance level of 0.001
Statistical Analysis 24: Comparison: Low Dose of Hydrocortisone vs High Dose of Hydrocortisone; Digit span backward - Working memory; Test type: Superiority or Other; p = 0.632, Wilcoxon (Mann-Whitney) — A Bonferroni correction for multiple comparisons was applied, resulting in a significance level of 0.001
Statistical Analysis 25: Comparison: Low Dose of Hydrocortisone vs High Dose of Hydrocortisone; Trail Making Test - Time condition A; Test type: Superiority or Other; p = 0.512, Wilcoxon (Mann-Whitney) — A Bonferroni correction for multiple comparisons was applied, resulting in a significance level of 0.001
Statistical Analysis 26: Comparison: Low Dose of Hydrocortisone vs High Dose of Hydrocortisone; Trail Making Test - Time condition B; Test type: Superiority or Other; p = 0.861, Wilcoxon (Mann-Whitney) — A Bonferroni correction for multiple comparisons was applied, resulting in a significance level of 0.001
Statistical Analysis 27: Comparison: Low Dose of Hydrocortisone vs High Dose of Hydrocortisone; Trail Making Test - Condition B/A; Test type: Superiority or Other; p = 0.958, Wilcoxon (Mann-Whitney) — A Bonferroni correction for multiple comparisons was applied, resulting in a significance level of 0.001
Statistical Analysis 28: Comparison: Low Dose of Hydrocortisone vs High Dose of Hydrocortisone; Social cognition; Test type: Superiority or Other; p = 0.819, Wilcoxon (Mann-Whitney) — A Bonferroni correction for multiple comparisons was applied, resulting in a significance level of 0.001

2. Secondary Outcome: Change in Quality of Life After 10 Weeks of Treatment With a Low Dose of Hydrocortisone Compared to 10 Weeks of Treatment With a High Dose of Hydrocortisone.
Description: Quality of life questionnaires have to be filled in by the participant at his/her home place and have to be returned by post.
Time Frame: as for outcome 1
Reporting Status: Not Posted

3. Secondary Outcome: Change in Metabolic Profile After 10 Weeks of Treatment With a Low Dose of Hydrocortisone Compared to 10 Weeks of Treatment With a High Dose of Hydrocortisone.
Description: Cardiovascular and metabolic risk factors, (pituitary) hormones and bone markers.
Time Frame: as for outcome 1
Reporting Status: Not Posted

4. Secondary Outcome: Change in Somatosensation After 10 Weeks of Treatment With a Low Dose of Hydrocortisone Compared to 10 Weeks of Treatment With a High Dose of Hydrocortisone.
Description: Measures of somatosensation: the mechanical detection threshold, the mechanical pain threshold, mechanical pain sensitivity, dynamic mechanical allodynia, wind up ratio and the pressure pain threshold.
Time Frame: as for outcome 1
Reporting Status: Not Posted

5. Secondary Outcome: Change in Perceived Common Somatic Complaints After 10 Weeks of Treatment With a Low Dose of Hydrocortisone Compared to 10 Weeks of Treatment With a High Dose of Hydrocortisone.
Description: The patients report common somatic complaints by filling in structured daily diaries.
Time Frame: during treatment period 1 (that is from week 1 to week 10 from baseline) and during treatment period 2 (that is from week 11 to week 20 from baseline).
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 4 weeks run in phase (if applicable) + 10 weeks (treatment period 1) + 10 weeks (treatment period 2)
Description: On testdays patients were questioned to report any adverse events. Furthermore, in week 5 and week 15 of the treatment period, patients were asked if any adverse events happened. In between these assessments patients were able to report any adverse events when necessary.
Groups:
- Low Dose of HC: Administration of a low dose of hydrocortisone (0.2-0.3 mg/kg body weight) for 10 weeks
- High Dose of HC: Administration of a high dose of hydrocortisone (0.4-0.6 mg/kg body weight) for 10 weeks
Arm/Group | Low Dose of HC | High Dose of HC
Serious Adverse Events (participants affected / at risk) | 1/58 | 1/55
Other Adverse Events (participants affected / at risk) | 20/58 | 13/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose of HC (N=58) | High Dose of HC (N=55)
Influenza A infection (Infections and infestations) | 1 (1) | 0 (0)
Minor stroke left cerebral hemisphere (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose of HC (N=58) | High Dose of HC (N=55)
Influenza (Infections and infestations) | 2 (2) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Tiredness (General disorders) | 3 (3) | 1 (1)
Joint pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Allergic reaction to Ibuprofen (Immune system disorders) | 0 (0) | 1 (1)
Progressive depression (Psychiatric disorders) | 1 (1) | 0 (0)
Dizziness (General disorders) | 1 (1) | 1 (1)
Headache (General disorders) | 1 (1) | 0 (0)
Cystitis (Renal and urinary disorders) | 1 (1) | 0 (0)
Stiffness in joints (General disorders) | 1 (1) | 0 (0)
Gasteroenteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cardiac catheterisation (Cardiac disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Herpes Zoster (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Nausea (General disorders) | 1 (1) | 1 (1)
Broken arm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Motorcycle accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Red spots in face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Diplopia with operative correction (Eye disorders) | 0 (0) | 1 (1)
Acne on back and forehead (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Fall from a horse (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes